CLINICAL TRIAL: NCT05122741
Title: Modulation of the WNT/Beta-Catenin Pathway in Patients With Acute Myocardial Infarction
Brief Title: Modulation of Fibrosis-inducing Pathways in Acute Myocardial Infarction
Acronym: BETA-MI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Messina (Other)
Collaborators: Natasha Irrera (Unknown); Gianluca Di Bella (Unknown); Antonio Micari (Unknown); Roberto Licordari (Unknown)
Responsible Party: Principal Investigator, Francesco Costa, Doctor, University of Messina
Other Study IDs: Cardio1
Record Dates: First submitted 2021-09-28; First posted 2021-11-17 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Myocardial Infarction; Myocardial Fibrosis; Myocardial Remodeling, Ventricular
Keywords: Myocardial Infarction; Beta-Catenin; WNT Signaling pathway; Adenosine systems; Dual Antiplatelet Therapy; Ticagrelor; Prasugrel; Myocardial Fibrosis; Clopidogrel
MeSH Terms: conditions — Myocardial Infarction; Ventricular Remodeling | interventions — Aspirin; 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine; Clopidogrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 45 Days
Biospecimen Retention: Samples Without DNA — Blood samples will be used to study:
  * serum concentrations of Adenosine, Beta-Catenin, cAMP
  * expression mRNAs encoding for Beta-Catenin.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Myocardial Infarction: 40 patients with clinical presentation of acute myocardial infarction undergoing primary percutaneous coronary intervention and eligible for dual antiplatelet therapy (DAPT) with either prasugrel or ticagrelor on top of aspirin.
  Interventions: Drug: P2Y12 Potent Inhibitor + Aspirin for STEMI patients
- Chronic Coronary Syndrome: 10 patients with stable coronary artery disease with an indication, according to current guidelines, to percutaneous coronary intervention and subsequent DAPT with aspirin and clopidogrel.
  Interventions: Drug: Clopidogrel + Aspirin for CCS patients

INTERVENTIONS:
Drug: P2Y12 Potent Inhibitor + Aspirin for STEMI patients — Patients will undergo primary percutaneous coronary intervention and DAPT with potent P2Y12 inhibitor (ticagrelor or prasugrel + aspirin)
  Other Names: DAPT with Potent P2Y12i
  Groups: Acute Myocardial Infarction
Drug: Clopidogrel + Aspirin for CCS patients — Patients will undergo elective percutaneous coronary intervention and DAPT with non-potent P2Y12 inhibitor (clopidogrel + aspirin)
  Other Names: DAPT with Clopidogrel
  Groups: Chronic Coronary Syndrome

SUMMARY:
This is a single-center, prospective, observational controlled cohort study designed to describe the role of WNT/B-catenin signaling and adenosine system after an acute myocardial infarction, correlating it with clinical markers of fibrosis/remodeling (primary objective). The modulation of the aforementioned molecular patterns will also be evaluated in light of the type of P2Y12 inhibitor implemented (ticagrelor or prasugrel) to identify variations in response (secondary objective).

DETAILED DESCRIPTION:
A total of 50 patients will be enrolled in the study, 40 with clinical presentation of acute myocardial infarction and eligible for treatment with either prasugrel or ticagrelor, and a control cohort of 10 patients with stable coronary artery disease, matched for age, sex and major risk factors, and with no history of prior myocardial infarction.

The study has been approved by the local ethics committee on 22/09/2021. Pre-enrollment screening will start from 01/11/2021. Blood samples will be obtained at 5 time-points: before and immediately after coronary revascularization (PCI) through the arterial introducer, and in the ward / clinic at a distance of 3, 5 days and 45±15 days from the procedure during normal routine examinations.

These will be used to study the expression of messenger RNA encoding for beta-catenin and to dose concentrations of beta-catenin, adenosine and cyclic adenosine monophosphate (cAMP) on serum. The extraction of RNA from blood samples will be carried out with a Real-time PCR method and the determination of molecules using ELISA colorimetric method, using specific kits.

Clinical-laboratory markers of left ventricular remodeling such as NT-proBNP, hsTnT, C-reactive protein, CK-MB, 12-lead ECG, transthoracic echocardiogram and cardiac magnetic resonance imaging, will be evaluated during hospitalization (at 3 and 5 days) and at the control visit (at 45 ± 15 days) as per standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ST segment elevation acute myocardial infarction undergoing coronary angiography and interventional treatment.*

  * Patients with chronic coronary syndrome matched by age, sex and risk factors will also be screened and included as per study design.
* Patients with an indication to potent P2Y12 inhibitor therapy (i.e. ticagrelor or prasugrel) for acute myocardial infarction.
* Population equally amenable to ticagrelor or prasugrel therapy according to the italian drug instruction of use (IFU)

Exclusion Criteria:

* Patients with a poor prognosis (less than 12 months)
* Patients admitted with cardiogenic shock or advanced cardiac failure (NYHA 4)
* Patients pre-treated before coronary angiography or in chronic therapy with a P2Y12 inhibitor
* Patients undergoing a medical only approach without percutaneous myocardial revascularization
* Patients undergoing surgical coronary revascularization
* Patients with prior history of myocardial infarction or prior coronary revascularization.
* Patients with contraindications or intolerance to antiplatelet therapy (ticagrelor, prasugrel, clopidogrel or cardioaspirin)
* Patients scheduled for a treatment with with cangrelor or GPIIb/IIIa inhibitors
* Patients with active bleeding at the time of inclusion
* Hemorrhagic diathesis
* Confirmed history of renal failure with glomerular filtration rate of <30ml/min
* Severe hepatopathy
* Patients treated or scheduled for treatment with oral anticoagulant therapy
* Active cancer or diagnosis any proliferative disease within 5 years.
* Prior TIA or stroke (ischemic or hemorrhagic)
* Age >75 years
* Weight <60kg

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients planned to undergo percutaneous coronary revascularization. A total of 50 patients will be enrolled in the study, 40 with clinical presentation of acute myocardial infarction with an indication for primary percutaneous coronary intervention and eligible for treatment with either prasugrel or ticagrelor, and a control cohort of 10 patients with stable coronary artery disease and no history of prior myocardial infarction who are not indicated for treatment with potent P2Y12 inhibitors.
  To ensure comparability the study and control groups, the control cohort will be matched to exclude a potential confounder effect of age, sex and other established risk factors.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between WNT/B-catenin levels and NTproBNP in patients presenting with acute myocardial infarction | Measured at 5 days after PCI
  NTproBNP as per center standard dosing
Correlation between WNT/B-catenin levels and and left ventricular ejection fraction in patients presenting with acute myocardial infarction | Measured at 5 days after PCI
  Left ventricular ejection fraction will be measured with transthoracic Echocardiography at the specified timepoint
Correlation between WNT/B-catenin levels and and extent of myocardial necrosis in patients presenting with acute myocardial infarction | Measured at 5 days after PCI
  Extent of myocardial necrosis will be measured with Carciac Magnetic Resonance Imaging at the specified timepoint
Correlation between in hospital WNT/B-catenin levels and NTproBNP at follow-up in patients presenting with acute myocardial infarction | Measured at 45 day after PCI
  NTproBNP as per center standard dosing
Correlation between in-hospital WNT/B-catenin levels and left ventricular ejection fraction at follow-up in patients presenting with acute myocardial infarction | Measured at 45 day after PCI
  Left ventricular ejection fraction will be measured with transthoracic Echocardiography at the specified timepoint
Correlation between in-hospital WNT/B-catenin levels and extent of myocardial fibrosis at follow-up in patients presenting with acute myocardial infarction | Measured at 45 day after PCI
  Extent of myocardial fibrosis will be measured with Carciac Magnetic Resonance Imaging at the specified timepoint

SECONDARY OUTCOMES:
Differences in WNT/B-catenin levels according to clinical presentation | At baseline, 3, 5 and 45 day after PCI
  Differences in results of activation of these molecular pathways in patients presenting with acute myocardial infarction and those selected in the control group by age, sex and risk factor matching
Differences in WNT/B-catenin levels in patients treated with ticagrelor or prasugrel | At baseline, 3, 5 and 45 day after PCI
  Differences in results of activation of these molecular pathways in patients treated with ticagrelor or prasugrel presenting with acute myocardial infarction
Differences in WNT/B-catenin levels in patients treated with or without Sodium-glucose Cotransporter-2 (SGLT-2) inhibitors | At baseline, 3, 5 and 45 day after PCI
  Differences in results of activation of these molecular pathways in patients treated or not treated with Sodium-glucose Cotransporter-2 (SGLT-2) inhibitors after acute myocardial infarction

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Policlinico G. Martino, Messina, Italy

IPD SHARING:
Plan to Share IPD: Undecided